CLINICAL TRIAL: NCT07211308
Title: Open and Closed Loop Differential Target Multiplexed Spinal Cord Stimulation in Patients With Persistent Spinal Pain Syndrome Type II: a European Multicenter Cohort Study (ENDLESS)
Brief Title: Open and Closed Loop DTM SCS in Patients With PSPS Type 2: ENDLESS Study
Acronym: ENDLESS
Status: Not yet recruiting | Type: Observational
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Sponsor
Other Study IDs: ENDLESS
Record Dates: First submitted 2024-11-07; First posted 2025-10-07 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-09

CONDITIONS: Persistent Spinal Pain Syndrome Type 2; Failed Back Surgery Syndrome; Failed Neck Surgery Syndrome
MeSH Terms: conditions — Failed Back Surgery Syndrome | interventions — Spinal Cord Stimulation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: Spinal Cord Stimulation — Differential target multiplexed stimulation

SUMMARY:
Evaluation of the effectiveness of differential target multiplexed spinal cord stimulation for treatment of Persistent Spinal Pain Syndrome Type II (PSPS-T2). Identification of clinical effective parameters concerning frequency, pulse duration, amplitude and battery consumption/recharge frequency and safety evaluation.

ELIGIBILITY:
Inclusion Criteria:

* having chronic pain as a result of PSPS-T2 that exists for at least 6 months with at least moderate pain intensity (4 or higher measured on numeric rating scale (NRS) or 31mm or higher measured on visual analogue scale (VAS) for the dominant pain location.
* being offered treatment with DTM SCS
* being at least 18 years old

Exclusion Criteria:

* Expected inability of patients to properly operate the SCS system
* History of coagulation disorders, lupus erythematosus, diabetic neuropathy
* Active malignancy
* Addiction to drugs and/or alcohol (more than 5 units /day)
* Evidence of an active disruptive psychiatric disorder or other known condition significant enough to impact perception of pain, compliance to intervention and/or ability to complete questionnaires, as determined by the investigator
* Immune deficiency (e.g. HIV positive, immunosuppressiva)
* Life expectancy < 1 year
* Local infection or other skin disorder at site of incision
* Pregnancy
* Other implanted active medical device

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Persistent Spinal Pain Syndrome type 2 (PSPS-T2), who will receive treatment with differential target multiplexed (DTM) SCS.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2028-01-01 (Estimated); Study Completion 2029-01-01 (Estimated)

PRIMARY OUTCOMES:
Overall pain intensity | The change between the baseline screening and the evaluation 1 month after DTM stimulation, 6 months and 12 months
  The primary effectiveness outcome measure is pain intensity measured with the Visual Analogue Scale (VAS), ranging from 0 (no pain) to 100 (maximal pain) in electronic format. Two scales will be presented for low back/neck pain and for leg/arm pain. Ecological momentary Assessment (EMA) will be used to collect pain intensity scores for VAS, whereby pain intensity is measured for multiple times per day for 1 week to reveal patterns of transient or fluctuating symptoms in the environment and context of the patients' lives, without a recall bias.

SECONDARY OUTCOMES:
Pain intensity for the lower back and leg pain or neck and arm pain component | The change between the baseline screening and the evaluation 1 month after DTM stimulation, 6 months and 12 months
  Pain intensity for the lower back and leg pain or neck and arm pain component will be assessed separately with the Numeric Rating Scale (0 to 10). Pain intensity for the last 7 days will be assessed in electronic format, with and without medication use.
Medication use | The change between the baseline screening and the evaluation 1 month after DTM stimulation, 6 months and 12 months
  Open question regarding the use of medication (collected through ecological momentary assessment for 1 week).
Negative affect | The change between the baseline screening and the evaluation 1 month after DTM stimulation, 6 months and 12 months
  Questions on a 9-point scale for negative affects, evaluated through ecological momentary assessment for 7 days.
Functional disability | The change between the baseline screening and the evaluation 1 month after DTM stimulation, 6 months and 12 months
  The Oswestry disability index (ODI; 0 to 100) or Neck disability index (NDI; 0 to 100) is used to measure functional disability due to abnormalities of the spine
Health related quality of life | The change between the baseline screening and the evaluation 1 month after DTM stimulation, 6 months and 12 months
  Health related quality of life, evaluated with the EuroQol with five dimensions and 5 levels
Patient global impression of change | Evaluated at 1 month, 6 months and 12 months of DTM SCS
  Patients will be asked to quantify the impression of change after treatment using the Patient Global Impression of Change scale (PGIC)
Clinical holistic responder status | The change between the baseline screening and the evaluation 1 month after DTM stimulation, 6 months and 12 months
  This is a composite measure for success, relying on the combination of the above questionnaires.
Work status | The change between the baseline screening and the evaluation 1 month after DTM stimulation, 6 months and 12 months
  Work status is evaluated with a self-designed questionnaire
Pain catastrophizing | The change between the baseline screening and the evaluation 1 month after DTM stimulation, 6 months and 12 months
  The Pain Catastrophizing Scale (PCS) will be used to measure the level of pain catastrophizing
Anxiety and Depression | The change between the baseline screening and the evaluation 1 month after DTM stimulation, 6 months and 12 months
  The hospital Anxiety and Depression Scale (HADS) will measure symptoms of anxiety and depression
Patient expectations concerning SCS | Evaluated at baseline visit
  Self-constructed open question to evaluate patient expectations about SCS
Patient unwanted stimulation awareness and satisfaction about the therapy | Evaluated at 1 month, 6 months and 12 months of DTM SCS
  investigated by self-reporting methods with 12 questions
Time spent in body postures | The data will be extracted from SCS implantation up to 1 month of SCS, from 1 month of SCS up to 6 months and from 6 months up to 12 months
  Based on the AdaptiveStim technology, the time spent in body postures can be recorded
(Serious) adverse events | Throughout study period, an average of 1 year
  Systematically recording all adverse events
Proportion of successful DTM trials | Evaluated after final SCS implantation
Technical IPG details (ECAPs etc.) | Registration at 1 month, 6 months and 12 months of DTM SCS
  Information from implantable pulse generators will be extracted.
DTM SCS stimulation parameters | Time Frame: Registration at 1 month, 6 months and 12 months of DTM SCS
  Information from implantable pulse generators will be extracted.
Battery consumption | Registration at 1 month, 6 months and 12 months of DTM SCS
  Information from implantable pulse generators will be extracted.
Prevalence of technical issues with regard to DTM SCS programming | Throughout study period, an average of 1 year
Actigraphy data | The change between the baseline screening and the evaluation 1 month after DTM stimulation, 6 months and 12 months
  A Garmin Venue series watch will be used to collect actigraphy data. Devices are worn for 7 consecutive days. This data will only be collected at Belgian sites.

CONTACTS AND LOCATIONS:
Locations (2):
- Belgium (2):
  - UZ Brussel, Brussels
  - Vitaz, Sint-Niklaas

IPD SHARING:
Plan to Share IPD: Undecided